CLINICAL TRIAL: NCT00983554
Title: Metabolic Effects of Testosterone Alone or in Combination With Dutasteride or Anastrazole in Obese Men
Brief Title: Metabolic Effects of Steroids in Obese Men
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of California, San Diego (Other)
Responsible Party: Karen L. Herbst, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DK65038 (completed)
Record Dates: First submitted 2009-09-22; First posted 2009-09-24 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Obesity; Insulin Resistance
Keywords: testosterone; insulin; obesity; aromatase; 5 alpha reductase
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Anastrozole; Testosterone; Dutasteride; LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (No Intervention)
- Anastrazole and Testosterone (Experimental)
  Interventions: Drug: Anastrazole; Drug: Testosterone; Drug: Dutasteride; Drug: GnRH antagonist
- Dutasteride and Testosterone (Experimental)
  Interventions: Drug: Testosterone; Drug: Dutasteride; Drug: GnRH antagonist
- Testosterone (Experimental)
  Interventions: Drug: Testosterone; Drug: Dutasteride; Drug: GnRH antagonist

INTERVENTIONS:
Drug: Anastrazole — Arimidex 1mg daily
  Arms: Anastrazole and Testosterone
Drug: Testosterone — Testim 10g daily
  Arms: Anastrazole and Testosterone; Dutasteride and Testosterone; Testosterone
Drug: Dutasteride — Avodart 2.5mg daily
  Arms: Anastrazole and Testosterone; Dutasteride and Testosterone; Testosterone
Drug: GnRH antagonist — Acyline 300 µg/kg subcutaneous injections every 2 weeks
  Arms: Anastrazole and Testosterone; Dutasteride and Testosterone; Testosterone

SUMMARY:
Subjects will be randomized into 4 study groups: 1. Placebo; 2. Anastrazole and Testosterone; 3. Dutasteride and Testosterone; and 4. Testosterone only. A 2 step euglycemic clamp, body composition by dual X-ray absorptiometry scan, hormone and lipid assays will be performed to monitor metabolic effects of each treatment group. We hypothesize that increasing testosterone levels would increase lean mass, decrease fat mass and improve insulin sensitivity. We further hypothesize that improvements in the metabolic profile would decrease with anastrazole and improve with dutasteride, given in conjunction with T administration.

ELIGIBILITY:
Inclusion Criteria:

* free T level in the lower 25% of the normal range or below
* BMI ≥30kg/m2
* waist circumference ≥100cm

Exclusion Criteria:

* pituitary tumors
* HIV infection
* Klinefelter's syndrome
* Kallman's syndrome
* uncontrolled hypertension
* diabetes
* congestive heart failure
* chronic lung disease
* acute coronary syndrome
* PSA >4µg/L
* aspartate aminotransferase (AST)> 3x upper limit of normal
* use of medications that might affect weight loss, muscle or bone metabolism or androgen metabolism, action or clearance.
* involvement in daily resistance training or high endurance exercise
* alcohol or drug dependence
* obstructive sleep apnea

Ages: 24 Years to 51 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2005-06; Primary Completion 2009-05 (Actual); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
insulin sensitivity | 14 weeks

SECONDARY OUTCOMES:
body composition | 14 weeks
lipid profile | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Herbst, PhD, MD, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - University of California, San Diego, San Diego, California
  - VA San Diego Healthcare System, San Diego, California

REFERENCES:
- [Background] Marin P, Holmang S, Gustafsson C, Jonsson L, Kvist H, Elander A, Eldh J, Sjostrom L, Holm G, Bjorntorp P. Androgen treatment of abdominally obese men. Obes Res. 1993 Jul;1(4):245-51. doi: 10.1002/j.1550-8528.1993.tb00618.x. PMID 16350577
- [Background] Marin P, Holmang S, Jonsson L, Sjostrom L, Kvist H, Holm G, Lindstedt G, Bjorntorp P. The effects of testosterone treatment on body composition and metabolism in middle-aged obese men. Int J Obes Relat Metab Disord. 1992 Dec;16(12):991-7. PMID 1335979
- [Background] DeFronzo RA, Tobin JD, Andres R. Glucose clamp technique: a method for quantifying insulin secretion and resistance. Am J Physiol. 1979 Sep;237(3):E214-23. doi: 10.1152/ajpendo.1979.237.3.E214. PMID 382871
- [Background] Kapoor D, Goodwin E, Channer KS, Jones TH. Testosterone replacement therapy improves insulin resistance, glycaemic control, visceral adiposity and hypercholesterolaemia in hypogonadal men with type 2 diabetes. Eur J Endocrinol. 2006 Jun;154(6):899-906. doi: 10.1530/eje.1.02166. PMID 16728551